CLINICAL TRIAL: NCT01406236
Title: Study of Access Site for Enhancement of PCI for Women (SAFE-PCI for Women)
Brief Title: SAFE-PCI for Women
Acronym: SAFE-PCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped for Statistical Futility. Low rate of bleeding events made it unlikely there would be statistical power to show a difference in the 2 arms.
Sponsor: Duke University (Other)
Collaborators: American College of Cardiology (Other); Abbott Medical Devices (Industry); Lilly USA (Unknown); Medtronic (Industry); Terumo Medical Corporation (Industry); The Medicines Company (Industry); Acist Medical Systems (Industry); Guerbet (Industry); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030109
Record Dates: First submitted 2011-06-20; First posted 2011-08-01 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Percutaneous Coronary Intervention; Ischemic Symptoms
Keywords: Female; urgent or elective percutaneous coronary intervention; PCI; diagnostic angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transradial PCI (Other)
  Interventions: Procedure: Transradial PCI
- Transfemoral PCI (Other)
  Interventions: Procedure: Transfemoral PCI

INTERVENTIONS:
Procedure: Transradial PCI — Transradial PCI
  Arms: Transradial PCI
Procedure: Transfemoral PCI — Transfemoral PCI
  Arms: Transfemoral PCI

SUMMARY:
The hypothesis of the SAFE-PCI for women trial is that, compared with transfemoral PCI, transradial PCI will result in a significant reduction in bleeding and vascular complications. The primary objective is to compare the efficacy and feasibility of the transradial approach to percutaneous coronary intervention (PCI) in women compared with the transfemoral approach.

This study is a multicenter, randomized, open-label active controlled study. Three thousand women undergoing urgent or elective PCI from at least 50 centers will be randomized to either transradial or transfemoral PCI. Patients who are enrolled at sites performing ad hoc PCI will be randomized before diagnostic angiography. A total of approximately 3000 women will be randomized to obtain a cohort of approximately 1800 patients undergoing PCI.

The Data Safety Monitoring Board has alerted us that the bleeding event rate overall in our trial is very low, making it unlikely that there will be statistical power to show a difference between the randomized arms in the SAFE PCI for Women study using the BARC bleeding definition per protocol. Based on this statistical futility, the DSMB has recommended stopping enrollment. They also noted, however, that as this is not based on any safety issues, and since there are a variety of key secondary endpoints (contrast and radiation exposure, quality of life) that are of clinical and scientific interest, the DSMB left it to the discretion of the Steering Committee to continue enrollment to meet sufficient power for these outcomes. On March 1, 2013, the Steering Committee met to discuss these issues and voted to continue enrollment until the planned sample size for the Quality of Life substudy was met (300 patients).

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to understand and sign an informed consent form
* Age ≥ 18 years
* Female patient undergoing urgent or elective PCI or undergoing diagnostic angiography to evaluate ischemic symptoms with the possibility of PCI

Exclusion Criteria:

* Peripheral arterial disease that prohibits vascular access
* Bilateral abnormal Barbeau tests
* Hemodialysis access (arteriovenous fistula or graft) in the arm to be used for PCI in case of assignment to radial approach (note that the opposite arm may be used for radial access in case a dialysis graft is present in one arm provided that the opposite arm has a normal Barbeau test)
* International normalized ratio (INR) ≥ 1.5 in a patient treated with oral vitamin K antagonists (i.e., warfarin).
* Receipt of oral Factor Xa or IIa inhibitors ≤ 24 hours prior to the procedure
* Planned staged PCI within 30 days of index procedure
* Valvular heart disease requiring valve surgery
* Planned right-heart catheterization
* Primary PCI for ST-segment elevation myocardial infarction
* Presence of bilateral internal mammary artery coronary bypass grafts
* Unable to provide informed consent
* Participation in any investigational drug or device study currently or within 30 days prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1787 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Composite of BARC Types 2, 3, and 5 bleeding or vascular complications. | From first arterial access post-randomization to 72 hours or hospital discharge, whichever occurs first.
Primary Feasibility Endpoint: Procedural failure, defined as inability to complete the procedure from the assigned vascular access site. | From first arterial access post-randomization to 72 hours or hospital discharge, whichever occurs first.

SECONDARY OUTCOMES:
Procedure Duration, total radiation dose and total contrast volume | 72 hours post randomization or hospital discharge (whichever occurs first)
  To determine the effect of transradial PCI on procedure time, total radiation dose, and total contrast volume.
Resource Use, patient preferences and quality of life | Baseline, 72 hours post randomization or hospital discharge (whichever occurs first), 30 day
  To determine the effect of transradial PCI on resource use, patient preferences, and quality of life.
30-day death, vascular complications, or repeat revascularization | 30 day
  To determine the effect of transradial PCI on 30-day death, vascular complications, or repeat revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil V Rao, MD, Principal Investigator — Duke University

REFERENCES:
- [Derived] Rymer JA, Kaltenbach LA, Kochar A, Hess CN, Gilchrist IC, Messenger JC, Harrington RA, Jolly SS, Jacobs AK, Abbott JD, Wojdyla DM, Krucoff MW, Rao SV. Comparison of Rates of Bleeding and Vascular Complications Before, During, and After Trial Enrollment in the SAFE-PCI Trial for Women. Circ Cardiovasc Interv. 2019 May;12(5):e007086. doi: 10.1161/CIRCINTERVENTIONS.118.007086. PMID 31014090
- [Derived] Rao SV, Hess CN, Barham B, Aberle LH, Anstrom KJ, Patel TB, Jorgensen JP, Mazzaferri EL Jr, Jolly SS, Jacobs A, Newby LK, Gibson CM, Kong DF, Mehran R, Waksman R, Gilchrist IC, McCourt BJ, Messenger JC, Peterson ED, Harrington RA, Krucoff MW. A registry-based randomized trial comparing radial and femoral approaches in women undergoing percutaneous coronary intervention: the SAFE-PCI for Women (Study of Access Site for Enhancement of PCI for Women) trial. JACC Cardiovasc Interv. 2014 Aug;7(8):857-67. doi: 10.1016/j.jcin.2014.04.007. PMID 25147030
- [Derived] Hess CN, Rao SV, Kong DF, Aberle LH, Anstrom KJ, Gibson CM, Gilchrist IC, Jacobs AK, Jolly SS, Mehran R, Messenger JC, Newby LK, Waksman R, Krucoff MW. Embedding a randomized clinical trial into an ongoing registry infrastructure: unique opportunities for efficiency in design of the Study of Access site For Enhancement of Percutaneous Coronary Intervention for Women (SAFE-PCI for Women). Am Heart J. 2013 Sep;166(3):421-8. doi: 10.1016/j.ahj.2013.06.013. Epub 2013 Jul 23. PMID 24016489